CLINICAL TRIAL: NCT00585221
Title: A Phase II Study Combining Targeted Therapy With Immunotherapy Using Imatinib Plus Peginterferon α-2b in Gastrointestinal Stromal Tumor (GIST) Patients
Brief Title: Study of Imatinib and Peginterferon α-2b in Gastrointestinal Stromal Tumor (GIST) Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI terminated at the recommendation of DSMC & IRB
Sponsor: University of Utah (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00022172
Record Dates: First submitted 2007-12-21; First posted 2008-01-03 (Estimated); Results first posted 2012-11-21 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Gastrointestinal Stromal Tumors; Cancer Brain; Solid Tumors
Keywords: Gastrointestinal stromal tumors; Imatinib; Peginterferon α-2b; Immunotherapy; Targeted therapy
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Brain Neoplasms | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All participants enrolled in the study.
  Interventions: Drug: Peginterferon-alpha 2b (PegIFNa2b);; Drug: Imatinib

INTERVENTIONS:
Drug: Peginterferon-alpha 2b (PegIFNa2b); — Treatment include PegIFNa2b high dose (3 mcg/kg/wk) X 4 doses and low dose (1.5 mcg/kg/wk) X 18 doses, followed by surgical evaluation to render pt disease free if possible.
  Other Names: Trade name: Peg-Intron
Drug: Imatinib — Continue imatinib until progression.
  Other Names: Trade name: gleevec

SUMMARY:
Imatinib (IM) has dramatically improved survival of gastrointestinal stromal tumors (GIST). However, most patients become resistant to IM in less than two years. This clinical trial combines targeted therapy (IM) with immunotherapy (peginterferon α-2b). Hypothesis: Apoptosis/necrosis of imatinib-sensitive GIST releases GIST-specific antigens in vivo while Peginterferon α-2b fulfills the role of cytokine signal (danger signal), this combination can induce effective innate and adaptive anti-GIST immunity, which can eradicate imatinib-resistant clones and GIST stem cells via recognition of common antigens shared with imatinib-sensitive GIST, leading to improved response rate and remission duration.

ELIGIBILITY:
1. Patients must be >18 years old.
2. Patients must have histologic evidence of GIST (Gastrointestinal Stromal Tumors).
3. If genotyping was not done, a paraffin block or 7 unstained slides or biopsy unstained slides is required for genotyping within one week of enrollment.
4. Stage I, II, and III patients are eligible if the primary tumor is 6 centimeter or larger. All stage IV (4) metastatic or recurrent GIST patients who are imatinib-naïve are eligible. For stage IV patients who had initial good response to imatinib and stopped imatinib for 10 months or longer. GIST patients who received imatinib as "adjuvant" treatment in the past, later developed a recurrence are eligible only if the DFS is > 6 months after completion of adjuvant imatinib.
5. Patients must have a Zubrod Performance Status of 0-1 or Karnofsky Performance Status >70%.
6. Patients must have a life expectancy of more than twelve months.
7. Patients must have negative serology tests for HIV (Human immunodeficiency virus). Hepatitis B, Hepatitis C, and ANA (antinuclear antibodies) titer have to be within 2 times of upper limit of normal within 28 days of enrollment. Patients must have no clinical rheumatoid arthritis (RA). RA criteria are as follows: 1) morning stiffness in and around joints lasting at least 1 hour before maximal improvement; 2) soft tissue swelling (arthritis) of 3 or more joint areas observed by a physician; 3) swelling (arthritis) of the proximal interphalangeal, metacarpophalangeal, or wrist joints; 4) symmetric swelling (arthritis); 5) rheumatoid nodules; 6) the presence of rheumatoid factor; and 7) radiographic erosions and/or periarticular osteopenia in hand and/or wrist joints.

   Criteria 1 through 4 must have been present for at least 6 weeks. RA is defined by the presence of 4 or more criteria. Patients must have normal thyroid function tests (1.5 times of upper and lower normal limit) including TSH (Thyroid-stimulating Hormone), and T4 (Thyroxine) within 4 weeks of enrollment.
8. Patients must have adequate liver function as evidenced by the following: total bilirubin, and AST (aspartate aminotransferase) < 2 times of institutional upper limit of normal assessed within 2 weeks of enrollment. If patient has extensive liver metastasis which is the main cause of abnormal liver function, this requirement does not apply. The Principal Investigator can use his or her clinical judgment.
9. Patients must have serum creatinine <2 miligrams/deciliter within 2 weeks of enrollment.
10. Patients must have WBC (white blood cells) > 3x109 /L, absolute neutrophil count (ANC) > 1.5 x 109 /L platelet count > 125 x 109 /L, hemoglobin > 11 within 2 weeks of enrollment.
11. Patients must have PT (prothrombin time), PTT (partial thromboplastin time) and INR (international normalized ratio) < institutional upper limit of normal within 4 weeks of enrollment.
12. Patients must have no history of malignancy other than atypical melanocytic hyperplasia, basal or squamous skin cancer or any in situ cancer, lobular carcinoma of the breast in situ, cervical cancer in situ, Clark I melanoma in situ or have been continuously disease free for 5 years prior to enrollment.
13. Patients may not have received chemotherapy within 30 days prior to enrollment.
14. Patients must have a negative serum pregnancy test if female of childbearing potential.
15. Patients must agree to use an accepted and effective method of contraception while on Pegintron and for a period of 18 months after completing or discontinuing Pegintron.
16. Patients may not have autoimmune disorder, or immunodeficiency.
17. Patients may not have undergone splenectomy or gastrectomy for any reason. Total gastrectomy usually results in poor tolerance to the recommended dose of Imatinib.
18. Patients cannot require antihistamines, non-steroidal anti-inflammatory drugs, or corticosteroids.
19. Patients may not have active ischemic heart disease or cerebrovascular disease, congestive heart failure (New York Heart Association class III or IV), or angina requiring ongoing medications. EKG (Electrocardiography) may not show acute ischemic changes or acute heart rhythm changes.
20. Patients cannot show a history of Central Nervous System demyelination, inflammatory disease or hereditary or acquired peripheral neuropathy greater than Grade 2.
21. Patients cannot have an ongoing psychiatric disorder, surgical condition, or medical condition requiring a treatment regimen that may interfere with the completion of this trial or the evaluation of safety and efficacy of the study compound. For any questions, please contact the study Principal Investigator.
22. Patients cannot be taking coumadin, lovenox or heparin for metallic heart valve or hypercoagulability.
23. Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.
24. In the opinion of the Principal Investigator the patient is eligible and a good candidate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lei Chen, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Chen LL, Chen X, Choi H, Sang H, Chen LC, Zhang H, Gouw L, Andtbacka RH, Chan BK, Rodesch CK, Jimenez A, Cano P, Jones KA, Oyedeji CO, Martins T, Hill HR, Schumacher J, Willmore C, Scaife CL, Ward JH, Morton K, Randall RL, Lazar AJ, Patel S, Trent JC, Frazier ML, Lin P, Jensen P, Benjamin RS. Exploiting antitumor immunity to overcome relapse and improve remission duration. Cancer Immunol Immunother. 2012 Jul;61(7):1113-24. doi: 10.1007/s00262-011-1185-1. Epub 2011 Dec 24. PMID 22198309

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All participants enrolled.
Period: Overall Study
Arm/Group | All Patients
Started | 8
Completed | 0
Not Completed | 8
Not completed — Protocol Violation | 8

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.875 (17.97)
Gender [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Decrease in Tumor Size.
Description: Response rate is measured by PET-CT scan (a decrease in standardized uptake value (SUV) by 25%), Response Evaluation Criteria in Solid Tumors (RECIST), and Choi criteria (10% decrease in tumor size or a 15% decrease in tumor density on contrast-enhanced CT, computed tomography, scan).
Time Frame: 18 months
Arm/Group | All Patients
Number analyzed (Participants) | 0

2. Primary Outcome: Time to Progression (TTP).
Time Frame: two years
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: Study procedures were not completed on any of the 8 participants. There are no AEs to report.
Groups:
- All Enrolled: All participants enrolled
Arm/Group | All Enrolled
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No